CLINICAL TRIAL: NCT06593678
Title: Telerehabilitation in Cancer Patients: Optimization of Prehabilitation and Rehabilitation Following Colorectal Resection. A Randomized Clinical Trial
Brief Title: Telerehabilitation in Cancer Patients: Optimization of Prehabilitation and Rehabilitation Following Colorectal Resection
Acronym: CCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Universidad de Zaragoza (Other); Universidad San Jorge (Other); Hospital Royo Villanova de Zaragoza (Unknown)
Responsible Party: Principal Investigator, Sandra Calvo Carrión, PhD, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZ-USJ-CCR
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Telerehabilitation; Physical Therapy
Keywords: Colorectal Cancer; Telerehabilitation; Physical Therapy; Functional Recovery; Multimodal program; Quality of life; Psychosocial factors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, sigle-blind randomized clinical trial with two parallel interventions
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group. Asynchronous telerehabilitation (Experimental): Receive a home-based rehabilitation program via an asynchronous digital telerehabilitation platform.
  Interventions: Other: Telerehabilitation Program
- Control Group. Booklet-based rehabilitation (Active Comparator): Receive a booklet-based rehabilitation program at home through a detailed printed guide (explanatory booklet).
  Interventions: Other: Booklet-based rehabilitation program

INTERVENTIONS:
Other: Telerehabilitation Program — Participants in the intervention group will receive a home-based rehabilitation program delivered via an asynchronous digital telerehabilitation platform. The multimodal program is accessible at online platform and it is composed for therapeutic exercises, including aerobic and strength training exercises, aimed at improving functional capacity and quality of life before and after colorectal cancer surgery.
  Other Names: Asynchronous Digital Rehabilitation
  Arms: Intervention Group. Asynchronous telerehabilitation
Other: Booklet-based rehabilitation program — Participants in the control group will receive a booklet-based rehabilitation program at home, provided through a detailed printed guide (explanatory booklet). This guide includes instructions in pictures and text for the multimodal program. It is composed for therapeutic exercises, including aerobic and strength training exercises, aimed at improving functional capacity and quality of life before and after colorectal cancer surgery.
  Other Names: Printed Guide Rehabilitation
  Arms: Control Group. Booklet-based rehabilitation

SUMMARY:
This study, titled: Telerehabilitation in Oncology Patients: Optimization of Prehabilitation and Rehabilitation Post-Colorectal Resection. Is a randomized clinical trial conducted at the Royo Villanova Hospital in Zaragoza, Spain. It aims to evaluate the effectiveness of a tele-rehabilitation program in enhancing functional capacity and quality of life for patients undergoing colorectal cancer surgery. Colorectal cancer (CRC) is a highly prevalent malignant tumor that significantly impacts global health and patients' quality of life, particularly after surgery. Prehabilitation and postoperative rehabilitation are crucial for recovery, and telerehabilitation offers a promising alternative to improve outcomes in CRC patients.

DETAILED DESCRIPTION:
Study Background and Rationale: Colorectal cancer (CRC) is one of the most prevalent malignant tumors worldwide and a leading cause of cancer-related deaths. Despite advancements in surgical and oncological treatments, patients often experience significant postoperative complications and a decline in their quality of life. Prehabilitation, which aims to enhance a patient's functional capacity before surgery, has been identified as a promising approach to improve postoperative outcomes. However, traditional rehabilitation programs are often limited by patient adherence, accessibility, and the availability of resources, especially for those living in rural or underserved areas.

Objective: The primary objective of this study is to determine whether a 2-week prehabilitation and 4-week post-surgical rehabilitation program delivered via asynchronous telerehabilitation software can improve the functional capacity of patients undergoing colorectal cancer surgery, as measured by the Six Minute Walking Test (6MWT). Secondary objectives include assessing changes in body composition, muscle strength, pulmonary capacity, postoperative complications, psychosocial factors (such as quality of life, anxiety, depression, and sleep quality), adherence to the treatment, patient acceptance of the treatment, and the usability of the telerehabilitation platform.

Study Design: This is a single-blind, parallel-group randomized clinical trial. Fifty-four patients scheduled for colorectal cancer surgery will be recruited and randomly assigned to either the control group, which will receive conventional rehabilitation through a booklet, or the intervention group, which will receive the same rehabilitation program through a digital telerehabilitation platform. Both groups will undergo a comprehensive rehabilitation program including therapeutic education, respiratory exercises, aerobic exercises, and strength training.

Methodology: Patients will be assessed at five time points: pre-intervention, the day before surgery, 21 days post-surgery, 50 days post-surgery, and 3-month follow-up. The telerehabilitation platform will allow patients to access exercise videos and therapeutic content asynchronously, with the ability to communicate with their physiotherapists through the platform for guidance and support. The booklet will allow patients to access the program through pictures and text.

Clinical implications: Telerehabilitation represents an innovative approach to overcoming barriers associated with conventional rehabilitation, particularly in improving accessibility for patients in remote areas. By demonstrating the clinical efficacy of telerehabilitation, this study aims to contribute to the optimization of rehabilitation protocols for oncology patients and to provide a scalable model for integrating digital health solutions into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years.
* Participants who understand Spanish.
* Patients scheduled for colorectal cancer surgery at Royo Villanova Hospital, Zaragoza, Spain.
* Patients attending the first consultation in the General and Digestive Surgery Section under the supervision of Dr. Blas, head of surgery at Royo Villanova Hospital, Zaragoza, Spain.
* Participants with functional independence that allows them to perform walking and pulmonary function tests.
* Patients with a preoperative assessment score of I, II, or III on the American Society of Anesthesiologists (ASA) scale.
* Participants who agree to participate and sign the informed consent form.

Exclusion Criteria:

* Patients older than 80 years.
* Patients with a preoperative ASA score of IV.
* Patients with any injury, pathology, or inflammatory processes that make it impossible to practice exercise.
* Patients with central and/or peripheral neurological diseases that prevent them from following the rehabilitation program.
* Patients with unstable cardiac comorbidities such as arrhythmias, high blood pressure, angina pectoris, or other conditions that contraindicate moderate-intensity training.
* Patients diagnosed with a psychiatric disorder as confirmed by a psychiatrist.
* Patients without access to mobile internet or a computer with internet at home.
* Patients who score ≤ 24 on the Mini-Mental State Examination (MMSE).
* Individuals who are unable to follow oral and written instructions in Spanish.
* Patients who refuse to participate in the study or who have not signed the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity - Six Minute Walking Test (6MWT) | Functional capacity will be assessed at four time points: pre-intervention (T1), the day before surgery (T2), 21 days post-surgery (T3), and 50 days post-surgery (T4).
  The primary outcome is the improvement in functional capacity, which will be evaluated using the Six Minute Walking Test (6MWT). This test measures the maximum distance a patient can walk in six minutes along a flat, straight corridor under controlled conditions. The results provide an objective assessment of the patient's functional capacity, reflecting their ability to perform daily activities and their level of postoperative recovery.

SECONDARY OUTCOMES:
Pulmonary Capacity - Spirometry Assessments | Measured at pre-intervention (T1), the day before surgery (T2), 21 days post-surgery (T3), and 50 days post-surgery (T4).
  Evaluate improvements in pulmonary capacity using spirometry, with a specific focus on measuring Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1) through standardized spirometry techniques.. The aim is to determine whether the tele-rehabilitation program can enhance respiratory function as compared to the standard approach.
Upper Limb Muscle Strength - Hand Grip Test | Measured at pre-intervention (T1), the day before surgery (T2), 21 days post-surgery (T3), and 50 days post-surgery (T4).
  Evaluate the muscle strength of the upper limbs using the Hand Grip Test. This assessment will provide data on the effectiveness of the tele-rehabilitation program in enhancing upper limb muscle strength.
Lower Limb Muscle Strength - Sit to Stand Test | Measured at pre-intervention (T1), the day before surgery (T2), 21 days post-surgery (T3), and 50 days post-surgery (T4).
  Evaluate the muscle strength of the lower limbs using the Sit to Stand Test. This assessment will provide data on the effectiveness of the tele-rehabilitation program in enhancing lower limb muscle strength.
Body Composition - Bioelectrical Impedance Analysis and Waist-to-Hip Ratio | Measured at pre-intervention (T1), the day before surgery (T2), 21 days post-surgery (T3), and 50 days post-surgery (T4).
  Assess changes in body composition, including measurements taken via bioelectrical impedance analysis (BIA) and waist-to-hip ratio. This will help determine if the tele-rehabilitation program leads to significant improvements in body composition compared to the conventional rehabilitation program.
Postoperative Complications - Comprehensive Complication Index (CCI) | Evaluated 3 months post-surgery (T5).
  Assess the occurrence and severity of postoperative complications using the Comprehensive Complication Index (CCI). The CCI provides a cumulative score that reflects the overall burden of all complications, ranging from 0 (no complications) to 100 (death). This outcome measure aims to determine whether the tele-rehabilitation program effectively reduces the rate and severity of postoperative complications compared to the standard rehabilitation approach.
Quality of Life - EuroQol-5D (EQ-5D) | Assessed at pre-intervention (T1), 50 days post-surgery (T4) and 3 months post-surgery (T5).
  Assess the impact on quality of life using the EuroQol-5D (EQ-5D) instrument. The EQ-5D evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores range from -0.594 to 1, where higher scores indicate better quality of life.
Anxiety and Depression - Hospital Anxiety and Depression Scale (HADS) | Assessed at pre-intervention (T1), 50 days post-surgery (T4) and 3 months post-surgery (T5).
  Measure levels of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of two subscales: anxiety and depression, each ranging from 0 to 21. Higher scores indicate worse outcomes.
Psychological Adjustment - Mental Adjustment to Cancer Scale (MAC) | Assessed at pre-intervention (T1), 50 days post-surgery (T4) and 3 months post-surgery (T5).
  Evaluate psychological adjustment to cancer using the Mental Adjustment to Cancer Scale (MAC). The MAC includes subscales such as fighting spirit, helplessness/hopelessness, anxious preoccupation, fatalism, and avoidance. Scores vary by subscale, generally ranging from 0 to 32 for each subscale. Higher scores on positive subscales, such as fighting spirit, indicate better adjustment, while higher scores on negative subscales, such as helplessness/hopelessness, indicate worse adjustment.
Sleep Quality - Pittsburgh Sleep Quality Index (PSQI) | Assessed at pre-intervention (T1), 50 days post-surgery (T4) and 3 months post-surgery (T5).
  Assess sleep quality using the Pittsburgh Sleep Quality Index (PSQI). The PSQI measures seven components: sleep duration, sleep disturbances, sleep latency, daytime dysfunction, and more. Scores range from 0 to 21, with higher scores indicating worse sleep quality.
Adherence to the Tele-Rehabilitation Program | Monitored continuously throughout pre-intervention (T1) - the day before surgery (T2), 21 days post-surgery (T3) - 50 days post-surgery (T4).
  Evaluate compliance with the tele-rehabilitation protocol by tracking the percentage of prescribed sessions completed by participants. Compliance data will be recorded in treatment diaries and through the tele-rehabilitation platform. The compliance rate will be calculated as the proportion of completed sessions out of the total prescribed sessions.
Satisfaction with Tele-Rehabilitation Program | Monitored continuously throughout pre-intervention (T1) - the day before surgery (T2), 21 days post-surgery (T3) - 50 days post-surgery (T4).
  Assess participant satisfaction with the tele-rehabilitation program using a standardized satisfaction survey. The survey will be recorded on the tele-rehabilitation platform, and scores will range from 1 to 4, with higher scores indicating greater satisfaction.
Incremental Cost-Effectiveness Ratio (ICER) - Cost per QALY | Evaluated after 3 months post-surgery (T5).
  Assess the cost-effectiveness of the tele-rehabilitation program compared to conventional clinical practice by calculating the Incremental Cost-Effectiveness Ratio (ICER). The ICER is expressed in euros per Quality-Adjusted Life Year (QALY). This measure will provide insight into the additional cost per QALY gained with the tele-rehabilitation program.
Quality-Adjusted Life Years (QALYs) | Evaluated after 3 months post-surgery (T5).
  Evaluate the quality-adjusted life years (QALYs) gained through the tele-rehabilitation program compared to conventional clinical practice. The QALY is a measure of the value of health outcomes, combining both quantity and quality of life. Scores typically range from 0 (equivalent to death) to 1 (perfect health), with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Calvo, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Hospital Royo Villanova, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No